CLINICAL TRIAL: NCT01812148
Title: Survival of Peritoneal Mesothelioma After Cytoreductive Surgery and Hyperthermic Intra-peritoneal Chemotherapy (HIPEC)
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Julien Hubert, Dr, Maisonneuve-Rosemont Hospital
Other Study IDs: Maisonneuve Rosemont Hospital; 12112 (Registry Identifier: Research Ethic committee of Maisonneuve Rosemont Hospital)
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Peritoneal Mesotheliomas
Keywords: Peritoneal Mesotheliomas; hyperthermic intra-peritoneal chemotherapy (HIPEC); Oxaliplatin; Cytoreductive surgery; Oxaliplatin HIPEC
MeSH Terms: interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Peritoneal Mesotheliomas: Cytoreductive surgery and HIPEC
  Interventions: Procedure: Cytoreductive surgery and HIPEC

INTERVENTIONS:
Procedure: Cytoreductive surgery and HIPEC — Cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy (HIPEC) with Oxaliplatin as chemotherapeutic agent

SUMMARY:
Review of the investigators hospital experience in cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy (HIPEC) for peritoneal mesotheliomas, using Oxaliplatin as intraperitoneal chemotherapeutic agent.

DETAILED DESCRIPTION:
Observation of primary outcome:

* Overall Survival
* Disease-free survival

Influencing factors that will be observe:

* Sex
* Blood loss
* Time of surgery
* Number of resection and anastomosis
* Peritoneal Index (PI score)
* Cytoreductibility (CCR score)

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal mesothelioma

Exclusion Criteria:

* Non resectable disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering of peritoneal mesotheliomas undergoing cytoreductive surgery and HIPEC
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Disease-Free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Sideris, MD, Study Director — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada